CLINICAL TRIAL: NCT01780935
Title: A 24-month, Phase IIIb, Randomized, Double-masked, Multicenter Study Assessing the Efficacy and Safety of Two Treatment Regimens of 0.5 mg Ranibizumab Intravitreal Injections Guided by Functional and/or Anatomical Criteria, in Patients With Neovascular Age-related Macular Degeneration
Brief Title: Efficacy and Safety of Two Treatment Regimens of 0.5 mg Ranibizumab Intravitreal Injections Guided by Functional and/or Anatomical Criteria, in Patients With Neovascular Age-related Macular Degeneration
Acronym: OCTAVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRFB002A2405; 2011-004959-39 (EudraCT Number)
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Results first posted 2017-01-02 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RBZ 0.5 mg: VA only (Group I) (Experimental): RBZ 0.5 mg: Visual Acuity (VA) only (Group I) 0.5 mg intravitreal injections of ranibizumab with retreatment based on best-corrected visual acuity (BCVA) loss due to neovascular (wet) age-related macular degeneration (nAMD)
  Interventions: Drug: Ranibizumab
- RBZ 0.5 mg: VA and/or OCT (Group II) (Experimental): RBZ 0.5 mg: VA and/or OCT (Group II) 0.5 mg intravitreal injections of ranibizumab with retreatment based on best-corrected visual acuity (BCVA)loss due to neovascular (wet) age-related macular degeneration (nAMD) and/or signs of wet AMD disease activity on optical coherence tomography (OCT).
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injections of 0.5 mg Ranibizumab

SUMMARY:
This study will evaluate and compare two individualized ranibizumab treatment regimens in patients with neovascular (wet) AMD aiming to achieve and to maintain a maximum visual function benefit, while aiming to avoid unnecessary intravitreal injections.

The results will be used to generate further recommendations on functional and anatomical monitoring of the disease and timing of treatment administration for patients with neovascular AMD. In this context, the study will investigate the utility of optical coherence tomography (OCT) to aid retreatment decisions with ranibizumab.

DETAILED DESCRIPTION:
During the course of the study, the use of optical coherence tomography (OCT)-guided therapy became a standard of care accepted by health authorities and the ophthalmology community in the treatment of neovascular (wet) age-related macular degeneration (nAMD), Novartis decided on 08-Oct-2014 the early termination of the study. Therefore the 12-month cutoff date was not reached and the related analyses were not performed.

ELIGIBILITY:
Inclusion Criteria:

* Visual impairment predominantly due to neovascular age-related macular degeneration AMD
* Active, newly diagnosed, untreated CNV due to AMD
* CNV involving the center of the retina
* A qualifying vision score at study entry

Exclusion Criteria:

* Stroke or myocardial infarction less than 3 Months prior to study entry
* Active injection or inflammation of either eye at the time of study entry

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2013-06-03 (Actual); Primary Completion 2015-07-09 (Actual); Study Completion 2015-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (82):
- Argentina (2):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As
- Novartis Investigative Site, Vienna, Austria
- Canada (6):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Boisbriand, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- Colombia (2):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Bogotá, Cundinamarca
- Czechia (4):
  - Novartis Investigative Site, Olomouc, CZE
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Prague
- Finland (2):
  - Novartis Investigative Site, HUS
  - Novartis Investigative Site, Kuopio
- Novartis Investigative Site, Paris, France
- Germany (8):
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Regensburg
- Greece (4):
  - Novartis Investigative Site, Ampelokipoi, Athens
  - Novartis Investigative Site, Glyfada, Athens
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Ioannina
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (5):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Veszprém
  - Novartis Investigative Site, Zalaegerszeg
- Ireland (2):
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Waterford
- Italy (3):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Udine, UD
- Lithuania (2):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Vilnius
- Novartis Investigative Site, Mexico City, Mexico City, Mexico
- Netherlands (3):
  - Novartis Investigative Site, 's-Hertogenbosch
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Panama City, Panama
- Portugal (3):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Slovakia (5):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Nitra
  - Novartis Investigative Site, Trenčín
  - Novartis Investigative Site, Zvolen
  - Novartis Investigative Site, Žilina
- Spain (5):
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Linköping, Sweden
- Switzerland (4):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Novartis Investigative Site, Ankara, Turkey (Türkiye)
- United Kingdom (15):
  - Novartis Investigative Site, Frimley, Surrey
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Cheshire
  - Novartis Investigative Site, Derby
  - Novartis Investigative Site, Gloucester
  - Novartis Investigative Site, Great Yarmouth
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Rugby
  - Novartis Investigative Site, Southampton
  - Novartis Investigative Site, Wolverhampton
  - Novartis Investigative Site, York

REFERENCES:
- [Derived] Staurenghi G, Garweg JG, Gerendas BS, Macfadden W, Gekkiev B, Margaron P, Dunger-Baldauf C, Kolar P. Functional versus functional and anatomical criteria-guided ranibizumab treatment in patients with neovascular age-related macular degeneration - results from the randomized, phase IIIb OCTAVE study. BMC Ophthalmol. 2020 Jan 9;20(1):18. doi: 10.1186/s12886-019-1251-6. PMID 31918685

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II)
Started | 335 | 336
Safety Set | 334 | 336
Completed | 0 | 0
Not Completed | 335 | 336
Not completed — Admin problems due to early termination | 321 | 309
Not completed — Adverse Event | 2 | 4
Not completed — Death | 1 | 6
Not completed — Lost to Follow-up | 2 | 6
Not completed — Physician Decision | 1 | 1
Not completed — Protocol deviation | 0 | 1
Not completed — Patient withdrew consent | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II) | Total
Number analyzed (Participants) | 335 | 336 | 671
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.9 (7.86) | 75.3 (7.91) | 74.6 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213 | 194 | 407
  Male | 122 | 142 | 264

OUTCOME MEASURES:

1. Primary Outcome: Average Best-corrected Visual Acuity (BCVA) (Letters) Change up to Month 12
Description: Visual acuity (VA) was assessed during every study visit using best correction determined from protocol refraction. VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like VA testing charts at a testing distance of 4 meters. This outcome measure describes the difference between the Visual Acuity averaged up to Month 12 Level of VA (Letters) of the Study Eye.
Time Frame: up to Month 12
Population: Full Analysis Set (FAS) includes all randomized patients
Measure: Mean (Standard Deviation); unit: Letters correctly read
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II)
Number analyzed (Participants) | 335 | 336
Letters correctly read | 0.1 (6.79) | 1.0 (7.25)

2. Secondary Outcome: Change From Baseline in Visual Acuity (Letters) of the Study Eye up to Month 12
Description: Visual acuity (VA) was assessed using best correction determined from protocol refraction. VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like VA testing charts at a testing distance of 4 meters. This outcome measure describes the difference between the Visual Acuity averaged from Baseline to Month 12 Level of VA (Letters) of the Study Eye.
Time Frame: up to Month 12
Population: Full Analysis Set (FAS) includes all randomized patients
Measure: Mean (Standard Deviation); unit: letters correctly read
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II)
Number analyzed (Participants) | 335 | 336
letters correctly read | 6.7 (13.48) | 8.3 (13.53)

3. Secondary Outcome: Gain of Equal or More Than 1, 5, 10, or 15 Letters in Visual Acuity of the Study Eye From Baseline, at Month 12 and 24
Description: During the course of the study, the use of optical coherence tomography (OCT)-guided therapy became a standard of care accepted by health authorities and the ophthalmology community in the treatment of neovascular (wet) age-related macular degeneration (nAMD), Novartis decided on 08-Oct-2014 the early termination of the study. Therefore the 12-month cutoff date was not reached and the related analyses were not performed.
Time Frame: Baseline to Month 12 and 24
Population: Early termination of the study, therefore the 12-month cutoff date was not reached and the related analysis was not performed
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Loss of Less Than 5, 10, and 15 Letters in Visual Acuity in the Study Eye From Baseline, at Month 12 and 24
Description: as for outcome 3
Time Frame: Baseline to Month 12 and 24
Population: as for outcome 3
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Visual Acuity of 73 Letters or More in the Study Eye at Month 12 and 24
Description: as for outcome 3
Time Frame: Month 12 and 24
Population: as for outcome 3
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Average Visual Acuity Change From Month 3 to Month 4 Through Month 24 in the Study Eye
Description: as for outcome 3
Time Frame: Month 3 to Month 24
Population: as for outcome 3
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Average Visual Acuity Change From Baseline to Month 1 Through Month 12 and 24 in the Study Eye
Description: as for outcome 3
Time Frame: Baseline to Month 12 and 24
Population: as for outcome 3
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Central Sub-Field Thickness (CSFT) and Central Sub-Field Volume (CSFV) of the Study Eye Over Time
Description: as for outcome 3
Time Frame: Baseline to Month 12 and 24
Population: as for outcome 3
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Dry Retina in the Study Eye on OCT at Month 12 and 24
Description: as for outcome 3
Time Frame: Month 12 and 24
Population: as for outcome 3
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Lesion Size and Morphology Based on Fluorescein Angiography at Month 12 and 24
Description: as for outcome 3
Time Frame: Baseline to Month 12 and 24
Population: as for outcome 3
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Treatment Patterns Over Time in Both Treatment Arms
Description: as for outcome 3
Time Frame: Baseline to Month 12 and 24
Population: as for outcome 3
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Functioning Questionnaire (NEI-VFQ-25) Scores Over Time
Description: as for outcome 3
Time Frame: Baseline to Month 12 and 24
Population: as for outcome 3
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Frequency and Severity of Ocular and Non-ocular Adverse Events Over Time
Description: as for outcome 3
Time Frame: Screening to Month 12 and 24
Population: as for outcome 3
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | RBZ 0.5 mg: VA Only (Group I) | RBZ 0.5 mg: VA and/or OCT (Group II)
Serious Adverse Events (participants affected / at risk) | 30/334 | 45/336
Other Adverse Events (participants affected / at risk) | 111/334 | 105/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RBZ 0.5 mg: VA Only (Group I) (N=334) | RBZ 0.5 mg: VA and/or OCT (Group II) (N=336)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 3
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Choroidal haemorrhage (Study eye) (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Fellow untreated eye) (Eye disorders) | 1 | 0
Retinal artery embolism (Study eye) (Eye disorders) | 0 | 1
Visual acuity reduced (Study eye) (Eye disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Neutropenic sepsis (Infections and infestations) | 0 | 1
Otitis media chronic (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 3
Tracheobronchitis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 4
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Visual acuity tests abnormal (Study eye) (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Encephalitis post varicella (Study eye) (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Breast calcifications (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Thrombophlebitis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RBZ 0.5 mg: VA Only (Group I) (N=334) | RBZ 0.5 mg: VA and/or OCT (Group II) (N=336)
Choroidal neovascularisation (Fellow untreated eye) (Eye disorders) | 5 | 7
Conjunctival haemorrhage (Study eye) (Eye disorders) | 19 | 10
Dry eye (Fellow untreated eye) (Eye disorders) | 7 | 4
Dry eye (Study eye) (Eye disorders) | 10 | 7
Eye pain (Study eye) (Eye disorders) | 10 | 9
Neovascular age-related macular degeneration (Fellow untreated eye) (Eye disorders) | 7 | 7
Vitreous floaters (Study eye) (Eye disorders) | 6 | 8
Bronchitis (Infections and infestations) | 7 | 6
Influenza (Infections and infestations) | 15 | 15
Nasopharyngitis (Infections and infestations) | 24 | 11
Urinary tract infection (Infections and infestations) | 2 | 7
Intraocular pressure increased (Study eye) (Investigations) | 12 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Hypertension (Vascular disorders) | 18 | 15

LIMITATIONS AND CAVEATS:
Use of optical coherence tomography guided therapy in the treatment of neovascular age related macular degeneration became standard of care by HA & Ophth. community during the time this trial was conducted.Novartis terminated this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.